CLINICAL TRIAL: NCT04087473
Title: Plasma Molecular Profiling in ALK Inhibitor Resistant Non-Small Cell Lung Cancer
Brief Title: Plasma Molecular Profiling in ALK Inhibitor Resistant NSCLC
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Guardant Health AMEA, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: ATORG004
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer; ALK-Positive Lung Cancer
Keywords: ALK inhibitor (ALKi); NSCLC; Anaplastic lymphoma kinase (ALK) fusion oncogene NSCLC; Guardant360 assay; Next-Generation Sequencing (NGS) DNA sequencing test; Cell-free circulating tumor DNA (ctDNA); Plasma profiling; Blood-based assay; Mutational testing; 74 genetic alterations (point mutations, copy number variants, fusions, insertions, deletions); ALK resistance mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15-20mL of plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prior 2nd generation ALKi
- Prior 1st and 2nd generation ALKi

SUMMARY:
The investigators plan to understand a comprehensive molecular profiling via the plasma, with the primary aim of using this form on analysis to guide subsequent treatment selection. This study will provide a better understanding of ALK resistance in the treatment of Asian lung cancers and allow for improved clinical outcomes by 'matching' the secondary mutations to an ALK inhibitor which would allow for the greatest coverage ultimately leading to lasting duration of response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced ALK fusion oncogene positive lung adenocarcinoma that have progressed after 1-2 ALK inhibitors, with at least one prior line of 2nd generation ALKi (i.e. Ceritinib, Alectinib, Brigatinib or Ensartinib)
* The availability of sufficient plasma
* Age ≥ 21 years
* WHO performance status ≤ 2
* Life expectancy of ≥ 21 weeks
* Patients should have adequate organ function for potential consideration into clinical trials (routine blood tests are valid within 14 days before enrollment):

  1. Adequate bone marrow function as shown by: ANC ≥ 1.0x10^9/L, Platelets ≥ 75x10^9/L, Hb ≥ 7.5 g/dL
  2. Alanine aminotransferase (ALT) and aspirate aminotransferase (AST) normal range (or ≤ 3.0xULN if liver metastases are present)
* Willing to provide signed informed consent
* Patients whom do not fulfill the above criteria may be discussed on a case-by-case basis within the study team, for potential enrolment

Exclusion Criteria:

* Received more than 2 prior ALK inhibitors (ALKi)
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment inclusive but not limited to surgery and radiation. Stable/ tailing doses of corticosteroids is permitted

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two cohorts will be enrolled, the first cohort will consist of patients that have received prior 2nd generation ALKi only, and the second cohort with patients that have received prior 1st and 2nd generation ALKi.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular profiling of plasma | 2 to 4 weeks after collection of plasma
  Profiling of the collected plasma samples at a molecular level to evaluate the molecular epidemiology of ALK fusion oncogene positive lung cancer

SECONDARY OUTCOMES:
Patient survival status | After molecular profiling has been completed, every few months up to 2 years
Subsequent patient treatment status | After molecular profiling has been completed, every few months up to 2 years
Clinical outcomes of the subsequent treatments the patients receive | After molecular profiling has been completed, every few months up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SW Tan, BSc, MBBS, PhD, Principal Investigator — National Cancer Centre of Singapore
Locations (5):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- National Cancer Center Singapore, Singapore, Singapore
- South Korea (2):
  - Asan Medical Centre, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No